CLINICAL TRIAL: NCT05233410
Title: Topical Ruxolitinib Evaluation in Chronic Hand Eczema Study 2 (TRuE-CHE2): A Phase 3, Double-Blind, Randomized, 16-Week, Vehicle Controlled, Efficacy and Safety Study of Ruxolitinib Cream Followed by an Open-Label Extension Period in Adults With Chronic Hand Eczema
Brief Title: Topical Ruxolitinib Evaluation in Chronic Hand Eczema Study 2
Acronym: TRuE-CHE2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision; no safety concerns
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-314
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Chronic Hand Eczema (CHE)
Keywords: eczema; hand eczema; dermatitis; skin disease; JAK inhibitor
MeSH Terms: conditions — Eczema; Dermatitis; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Participants will receive ruxolitinib cream (1.5%) or vehicle cream for 16 weeks, after which they will be offered the opportunity to receive ruxilitinib cream (1.5%) in the open-label treatment extension period for another 16 weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib (Experimental): Ruxolitinib cream 1.5% twice daily (BID) for 16 weeks followed by ruxolitinib cream 1.5% BID for an additional 16-week treatment extension period.
  Interventions: Drug: Ruxolitinib cream
- Vehicle (Placebo Comparator): Vehicle cream for 16 weeks followed by crossover to ruxolitinib cream 1.5% BID in a 16-week treatment extension period.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream is a topical formulation applied as a thin film to affected areas.
  Other Names: INCB18424 cream
  Arms: Ruxolitinib
Drug: Vehicle — Vehicle cream is a topical formulation applied as a thin film to affected areas.
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib cream in adult participants with diagnosis of chronic hand eczema (CHE) and moderate to severe disease activity (Investigator's Global Assessement (IGA) of CHE score 3 or 4).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chromic hand eczema (CHE) as defined by hand eczema (HE) lasting > 3 months or ≥ 2 flares within the previous 12 months.
* Screening and baseline IGA-CHE 3 or 4.
* Baseline CHE-related Itch NRS ≥ 4.
* Recent history (within the past 1 year of baseline) of inadequate response to treatment with topical corticosteroids (TCS), topical calcineurin inhibitors (TCI), or oral alitretinoin; or intolerance or contraindication to TCS or TCI or oral alitretinoin.
* Willingness to avoid pregnancy or fathering children based on the criteria below.

Exclusion Criteria:

* Known triggers for CHE (allergic or irritant, such as those identified by previous patch tests) cannot be avoided during the course of this study.
* Participants who have an unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to baseline.
* Participants with concurrent conditions and history of other diseases such as other active skin disease or infection on the hands; immunocompromised; chronic or acute infection requiring systemic treatments; active acute skin infection; other concomitant skin conditions that may interfere with study assessments or compromise participant safety; other types of eczema; chronic asthma requiring high dose of inhaled corticosteroids; current or history of hepatitis B or C virus infection.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Laboratory values outside of the protocol-defined criteria.
* Use of protocol-defined treatments within the indicated washout period before baseline.
* Psoralen ultraviolet A (PUVA) or ultraviolet B (UVB) therapy on the hands within 4 weeks before baseline.
* Pregnant or lactating participants, or those considering pregnancy during the period of their study participation.
* Further exclusion criteria apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2024-04-25 (Estimated); Study Completion 2024-09-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants achieving Investigator's Global Assessment-Chronic Hand Eczema Treatment Success (IGA-CHE-TS) | Week 16
  The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). IGA-CHE treatment success (IGA-CHE TS) is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from baseline.

SECONDARY OUTCOMES:
Percentage of Participants with a ≥ 4-point improvement in chronic hand eczema (CHE)-related Itch Numerical Rating Scale (NRS) score | Baseline to Week 16
  The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity and subjects will rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable) on a daily basis.
Percentage of Participants with a ≥ 2-point improvement in CHE-related Skin Pain NRS score | Baseline to Week 16
  The Pain NRS is a validated, self-reported, instrument for measurement of itch intensity and subjects will rate the intensity of their pain on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Change from baseline in the mTLSS (modified Total Lesion Symptom Score | Up to Week 32
  The mTLSS is a validated tool for assessing hand eczema. The scale quantifies the 7 features (erythema, scaling, hyperkeratosis/lichenification, vesiculation, oedema, fissures, and pruritus/pain) of HE (0 = none, 1 = mild, 2 = moderate, and 3 = severe).
Percentage of Participants achieving an IGA CHE-TS | Up to Week 32
  The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). IGA-CHE treatment success (IGA-CHE TS) is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from baseline.
Change from baseline in CHE-related Itch NRS score (weekly average) | Up to Week 32
  The Investigator's Global Assessment for chronic hand eczema (IGA-CHE) is an instrument used in clinical trials to rate the severity of the participant's global chronic hand eczema (CHE) and is based on a 5-point scale ranging from 0 (clear) to 4 (severe). IGA-CHE treatment success (IGA-CHE TS) is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from baseline.
Change from baseline in CHE-related Skin Pain NRS score (weekly average) | Up to Week 32
  The Pain NRS is a validated, self-reported, instrument for measurement of itch intensity and participants will rate the intensity of their pain on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Time to ≥ 4-point improvement in CHE-related Itch NRS score | Up to Week 32
  The Itch NRS is a validated, self-reported, instrument for measurement of itch intensity and participants will rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable) on a daily basis.
Time to ≥ 2-point improvement in CHE-related Skin Pain NRS score | Up to Week 32
  The Pain NRS is a validated, self-reported, instrument for measurement of itch intensity and participants will rate the intensity of their pain on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable) on a daily basis.
Percentage change in Hand Eczema Severity Index (HECSI) | Baseline to Week 16
  The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales.
Percentage of participants with HECSI-75 | Weeks 2, 8, 16, 32
  HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales.
Percentage of participants with HECSI-90 | Weeks 2, 8, 16, 32
  HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs (erythema, infiltration/papulation, vesicles, fissures, scaling, and oedema) and the extent of the lesions in each of the 5 hand regions (fingertips, fingers [except fingertips], palm of hands, back of hands, and wrists) by use of standard scales.
Mean Patient Global Impression of Change (PGIC) score | Up to Week 32
  The Patient Global Impression of Change (PGIC) is a participants' self-reporting measure that reflects their belief about the efficacy of treatment. The PGIC is a 7-point scale depicting a participant's rating of overall improvement of CHE and will be captured during site visits. It is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.
Percentage of participants with each score on the PGIC | Up to Week 32
  The PGIC is a participants' self-reporting measure that reflects their belief about the efficacy of treatment. The PGIC is a 7-point scale depicting a participant's rating of overall improvement of CHE and will be captured during site visits. It is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.
Percentage of participants with a score of either 1 or 2 on the PGIC | Up to Week 32
  The PGIC is a participants' self-reporting measure that reflects their belief about the efficacy of treatment. The PGIC is a 7-point scale depicting a participant's rating of overall improvement of CHE and will be captured during site visits. It is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.
Change from baseline in Dermatology Life Quality Index (DLQI) score | Up to Week 32
  The DLQI is a simple, 10 question (Q) validated quality-of-life questionnaire to measure how much the skin problem has affected the participant. It covers 6 domains including symptoms and feelings (Q1 and Q2), daily activities (Q3 and Q4), leisure (Q5 and Q6), work and school (Q7), personal relationships (Q8 and Q9), and treatment(Q10). The recall Period of this scale is over the last week. Response categories include 0-not at all, 1-a little, 2-a lot, and 3-very much, and unanswered or not relevant responses scored as 0. Scores range from 0 ("no impact on participant's life") to 30 ("extremely large effect on participant's life"), and a 4-point change from Baseline is considered as the minimal clinically important difference threshold. A negative change from Baseline indicates less impact of the skin problem on participant's life.
Change from baseline in EQ-5D-5L score | Up to Week 32
  EQ-5D-5L is a is a validated, self-administered, generic, utility questionnaire wherein participants will rate their current health state based on the following criteria: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change from baseline in Quality of Life in Hand Eczema Questionnaire (QOLHEQ) score | Up to Week 32
  The QOLHEQ is a validated instrument to assess disease specific Health Related Quality of Life (HRQOL) in patients suffering from hand eczema. The QOLHEQ is a disease specific instrument, thereby only assessing impairments caused by hand eczema. It consists out of 30 items which can be summarized according to four domains of HRQOL: Impairments because of (1) symptoms, (2) emotions, (3) limitations in functioning or (4) because of treatment and prevention.
Change from baseline in Working Limitations Questionnaire (WLQ) score | Up to Week 32
  The Work Limitations Questionnaire (WLQ) is a patient self-rated scale designed to assess on the-job impact of chronic health problems and/or treatment. The WLQ consists of 25 items in 4 dimensions: limitations handling time (5 items), physical work demands (6 items), mental interpersonal work demands (9 items), and output demands (5 items). Each item is rated on a 5- point scale from "All of the Time" (score 5) to "None of the Time" (score 0), or "Does Not Apply to My Job". The WLQ Productivity Loss Score is derived from the Global Productivity Index, which is calculated as a weighed sum of the 4 dimensions. Reduction in WLQ Productivity Loss score indicates less work limitation and represents the estimated percentage of productivity loss in the past two weeks due to presenteeism relative to a healthy benchmark sample. WLQ Productivity Loss Score ranges from 0% to 24.9%. Higher percent productivity loss reflects more severe work limitations.
Change from baseline in Work Productivity and Activity Impairment Questionnaire Specific Health Problem v2.0 in Chronic Hand Eczema (WPAI-SHP-CHE) | Up to week 32, followed by 30 days follow-up.
  The WPAI:SHP questionnaire assesses both work productivity through absenteeism (i.e., work time missed), presenteeism (i.e., impairment at work or reduced on-the-job effectiveness), and work productivity loss, as well as daily activity impairment (e.g., work around the house, shopping, exercising, childcare, studying) attributable to excess weight. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity. Negative numbers indicate improvement from baseline.
Number of Participants with Treatment Emergent Adverse Events (TEAE) | Up to 40 weeks
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Haq Nawaz, MD, Study Director — Incyte Corporation
Locations (38):
- United States (12):
  - University of Alabama Hospital, Birmingham, Alabama
  - Marvel Clinical Research LLC, Huntington Beach, California
  - Advanced RX Clin Research, Westminster, California
  - Advanced Rx Clinical Research, Westminster, California
  - Forcare Clinical Research, Tampa, Florida
  - Midwest Allergy Sinus Asthma, Sc, Springfield, Illinois
  - The Indiana Clinical Trials Center Ictc, Plainfield, Indiana
  - Delricht Research, Baton Rouge, Louisiana
  - Jubilee, Las Vegas, Nevada
  - Onsite Clinical Solutions, Llc Charlotte Central Office, Charlotte, North Carolina
  - Progressive Clinical Research, San Antonio, Texas
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin
- Bulgaria (5):
  - Medical Center Unimed Eood, Sevlievo
  - Dcc 'Alexandrovska', Eood, Sofia
  - Medical Center Hera Eood, Sofia
  - Dcc Xxviii, Sofia
  - Mc 'Synexus - Sofia', Eood, Sofia
- Canada (3):
  - Dr. Chih-Ho Hong Medical Inc., Surrey, British Columbia
  - Simcomed Health Ltd, Barrie, Ontario
  - Xlr8 Medical Research, Windsor, Ontario
- Czechia (3):
  - Fakultni Nemocnice U Sv. Anny V Brne, Brno
  - Clintrial SRO, Prague
  - Krajska Zdravotni A.S. - Masarykova Nemocnice V Usti Nad Labem O.Z., Ústí nad Labem
- Germany (9):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Derma-Study-Center Friedrichshafen Gmbh, Friedrichshafen
  - Dermatologikum Hamburg Gemeinschaftspraxis Gbr, Hamburg
  - Universitaetsklinikum Schleswig Holstein - Campus Luebeck, Lübeck
  - Gemeinschaftspraxis, Mahlow
  - Beldio Research Gmbh, Memmingen
  - Dermatologische Klinik Der Technischen Universitat Munchen, München
  - Klifos - Klinische Forschung Osnabrück, Osnabrück
- Etg Warszawa, Warsaw, Poland
- Spain (5):
  - Hospital General Universitario de Alicante, Alicante
  - Clinica Dermomedic, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital de Manises, Valencia

IPD SHARING:
Plan to Share IPD: No